CLINICAL TRIAL: NCT04492358
Title: Phase 2/3, Randomized, Open Study to Compare the Efficacy and Safety of Colchicine and Glucocorticoids Compared With the Standard of Treatment for Moderate/Severe COVID-19 in a Fragile and Vulnerable Population, Admitted to a Geriatric Hospital Unit or in a Transicional Care Center
Brief Title: Treatment for Moderate/Severe COVID-19 in a Fragile and Vulnerable Population, Admitted to a Geriatric Hospital Unit or in a Transicional Care Center
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No candidates for the recruitment
Sponsor: Maria Joyera Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Maria Joyera Rodríguez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-002462-14
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Prednisone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colchicine + prednisone (Experimental): Prednisone should be administered for 3 consecutive days (60 mg/d) together with colchicine (at doses of 0.5 to 1.5 mg/d, adjusted for weight and renal function) for 3 days and maintained for 14 days in total (0.5 mg/d).
  Interventions: Drug: Colchicine; Drug: Prednisone tablet
- Standard treatment (Active Comparator): The standard treatment used in each site will be administered to the patients assigned to the control group.
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: Colchicine — Colchicine: ideal dose of 0.3 mg/kg/day (or the dose that approximates that adjusted for age, weight and kidney function, and 0.5 mg and 1 mg tablets)
  Arms: colchicine + prednisone
Drug: Prednisone tablet — Prednisone 60 mg/day, in a single dose, during 3 days
  Arms: colchicine + prednisone
Drug: standard of care — The standard treatment used in each site will be administered to the patients assigned to the control group.
  Arms: Standard treatment

SUMMARY:
Study to compare the efficacy and safety of colchicine and glucocorticoids compared with the standard of treatment for moderate/severe COVID-19 in a fragile and vulnerable population, admitted to a geriatric hospital unit or in a transicional care center

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 65 years old and be admitted to the Geriatrics Unit of the Internal Medicine Service (Hospital Clínic de Barcelona) or to a transicional care center
2. Clinical diagnosis compatible with COVID-19 (in a favourable epidemiological context), with a disease considered moderate (grade 3-4) or severe (grade 5) according to the WHO 8-point ordinal scale for assessing clinical severity (https://www.who.int/publications/i/item/covid-19-therapeutic-trial-synopsis). This same scale will also be used to evaluate the evolution after the application of the corresponding treatment. Baseline clinical parameters will include the presentation of fever and any respiratory symptoms, both of upper respiratory tract and dyspnea, affecting the general state or gastrointestinal manifestations, since it is known that in elderly people the COVID-19 can present with atypical symptoms for a time that is difficult to determine, but it also tends to evolve to respiratory failure quickly and is associated with high mortality. For this reason, regardless of the time that has elapsed since the estimated onset of symptoms, patients with moderate - WHO grade 3, in whom the presence of fever, mild dyspnea or any gastrointestinal manifestation attributable to COVID-19 make an admission (in the case of hospital) and directed treatment (in all cases) advisable, will be candidates for inclusion in the study. Patients with moderate disease and oxygen requirements (WHO grade 4) and patients with severe pneumonia, but who can be managed initially with high flow oxygen therapy (WHO grade 5) may also be included in the study. The clinical diagnosis may be supported by radiological changes (via chest radiography, if available) suggestive of bilateral (established or incipient) pneumonia. At the time of diagnosis, biomarkers will also be collected, in an analysis that will include increased levels of C-reactive protein [PCR] and/or ferritin and microbiological confirmation of SARS-CoV-2.
3. Patients in whom the current clinical situation and the basal functional situation condition a prognosis that makes them consider a limited therapeutic ceiling, which includes the contraindication of applying more aggressive (e.g. non-invasive ventilation) or invasive measures (e.g. cardiopulmonary resuscitation or orotracheal intubation and mechanical ventilation), both in patients admitted to the Geriatric Unit (Hospital Clínic de Barcelona) and in those admitted to a transicional care center. The latter patients are also not considered for transfer to a third level hospital (according to the criteria of fragility, available on page 14 of the CatSalut action protocols (https://canalsalut.gencat.cat/web/.content/_A-Z/C/coronavirus-2019-ncov/material-divulgatiu/recull-protocol-pneumonia.pdf).
4. Patient with a general condition that allows him/her to take the medication orally, without risk of bronchial aspiration.
5. Acceptance by the patient or responsible family member to participate in the study (written consent).

Exclusion Criteria:

1. The clinical situation of an advanced or terminal illness, according to the clinical judgment of the doctor in charge and as defined by the Spanish Society for Palliative Care (SECPAL), which describes it as an advanced illness in an evolutionary and irreversible phase with multiple symptoms, emotional impact, loss of autonomy, with very little or no capacity to respond to specific treatment and with a life expectancy limited to weeks or months, in a context of progressive fragility (http://envejecimiento.csic.es/documentos/documentos/navarro-cuidadospaliativos-01.pdf).
2. Clinical status which is advanced and severe or in which the level of consciousness has deteriorated and the oral route of taking the medication is not safely tolerated (in the opinion of the doctor in charge)
3. Taking any of the drugs in the trial (colchicine or prednisone) chronically or intermittently in the 7 days prior to study inclusion.
4. Absolute contraindication to the use of the study medication, including hypersensitivity to the active substance or to any of its excipients, severe renal failure (glomerular filtration [GF] creatinine clearance or Clcr <30 ml/min) and patients undergoing haemodialysis, severe liver failure, severe gastrointestinal disorders, gastric ulcer or blood dyscrasias.
5. Concomitant treatment with macrolides (clarithromycin, erythromycin, telithromycin), antifungals (itraconazole, ketoconazole), cyclosporine and antivirals (lopinavir/ritonavir, indinavir, nelfinavir, saquinavir), all potent inhibitors of CYP3A4 (key cytochrome in the colchicine metabolism pathway).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients that a short cycle of steroids administered together with colchicine reduces mortality from COVID-19 | 28 days
  Number of patients that a short cycle of steroids (with prednisone 60 mg/d, in a single dose, for 3 consecutive days) administered together with colchicine (at doses of 0.5 to 1.5 mg/d, adjusted for weight and renal function, for 3 days and maintenance of 0.5 mg/d for 14 days in total) reduces mortality from COVID-19 in this population by at least 20%, compared to the approved standard treatment at participating centers.

SECONDARY OUTCOMES:
Number and grade of adverse events at group of colchicine and glucocorticoids throughout the treatment and in the two weeks following treatment | 28 days
  Number and grade of adverse events at group of colchicine and glucocorticoids throughout the treatment and in the two weeks following treatment according to the incidence of:
  * mild adverse event
  * serious adverse events
  * hypersensitivity (allergic) reactions of grade >=2
Percentage of patients who stop medication due to adverse events. | 28 days
  Percentage of patients who stop medication due to adverse events.
Severity of symptoms by COVID-19 in the two treatment arms | 28 days
  Severity of symptoms by COVID-19 in the two treatment arms (response to treatment to be assessed by overall survival at 28 days from the start of treatment).

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Centre Blauclínic Dolors Aleu, Barcelona
  - Hospital Clinic, Department of Internal Medicine, Barcelona
  - Clinica Sant Antoni, Barcelona

REFERENCES:
- [Derived] Hernandez-Rodriguez J, Duran-Sanclemente J, Prieto-Gonzalez S, Araujo O, Hospital-Vidal T, Casanovas G, Sapena V, Blanco JL, Lopez-Soto A; FRAGILE-COLCOVID19 Study Group. FRAGILE-COLCOVID19: A Clinical Trial Based on Early Administration of an Oral Combination of Colchicine and Prednisone in Elderly Patients with COVID-19 in Geriatric Facilities. Clin Drug Investig. 2022 Nov;42(11):949-964. doi: 10.1007/s40261-022-01201-2. Epub 2022 Sep 29. PMID 36173596